CLINICAL TRIAL: NCT04142125
Title: Combination Anti-thrombotic Treatment for Prevention of Recurrent Ischemic Stroke in Intracranial Atherosclerotic Disease: Protocol for a Pilot Randomized Trial
Brief Title: Combination Antithrombotic Treatment for Prevention of Recurrent Ischemic Stroke in Intracranial Atherosclerotic Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CATIS-ICAD
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke; Intracranial Atherosclerotic Disease
Keywords: Pilot study; Rivaroxaban; Factor Xa Inhibitors; Intracranial Atherosclerotic Disease
MeSH Terms: conditions — Ischemic Stroke | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Intervention Model Description: investigator-initiated, open-label, blinded endpoint assessment, controlled, randomized pilot trial (PROBE design)
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment of endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (riva + ASA) (Experimental): Rivaroxaban 2.5mg bid + aspirin 81mg qd
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet bid; Drug: Acetylsalicyclic acid 81 mg tablet qd
- Control (ASA alone) (Active Comparator): Aspirin 81 mg qd
  Interventions: Drug: Acetylsalicyclic acid 81 mg tablet qd

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet bid — Pts will receive rivaroxaban + aspirin
  Other Names: Xarelto
  Arms: Experimental (riva + ASA)
Drug: Acetylsalicyclic acid 81 mg tablet qd — Pts will receive ASA
  Other Names: Aspirin

SUMMARY:
CATIS-ICAD is a clinical pilot study in which patients who have had a recent ischemic stroke, that is a stroke caused by a blood clot or a narrowing of the blood vessels in the brain due to the build up of plaque, will be randomly assigned to receive either low-dose rivaroxaban + aspirin or aspirin alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Recent brain ischemia attributed to intracranial atherosclerotic stenosis of 30-99% as evidenced by CT or MR angiography, occurring between 7 to 100 days prior to randomization and consisting of either:

   1. a high-risk TIA defined as TIA with motor and/or speech involvement or
   2. an ischemic stroke
3. Written informed consent consistent with local regulations governing research in human subjects

Exclusion Criteria:

1. Indication for DAPT for > 90 days on guideline recommendations or investigator ́s judgment; e.g., cardiac stenting.
2. Indication for chronic anticoagulation based on guideline recommendations or investigator ́s judgment; e.g. patient with prosthetic mechanical valve, venous thromboembolism, hypercoagulable state
3. Atrial fibrillation or a history of atrial fibrillation
4. Intracranial arterial occlusion (e.g. 100% stenosis) responsible for the acute brain ischemia
5. Intracranial arterial stenosis secondary to causes other than atherosclerosis
6. Extracranial carotid artery disease ipsilateral to the qualifying brain ischemia with a plan for carotid revascularization
7. Intraluminal thrombus
8. Subdural hematoma within 12 months of randomization
9. Previous spontaneous hemorrhagic stroke (e.g. intracerebral or subarachnoid hemorrhage)
10. Traumatic brain hemorrhage within 1 month of randomization
11. Contraindication for MRI scan (e.g. pacemaker incompatible with MRI)
12. Advanced kidney disease (recent estimated GFR <30 ml per minute)
13. Modified Rankin Scale (mRS) >=4 at entry
14. Platelet count less than 100,000/mm3 at enrolment or other bleeding diathesis
15. Uncontrollable hypertension with systolic BP/ diastolic BP consistently above180/100mmHg after treatment
16. Known hypersensitivity to either ASA or rivaroxaban
17. Life expectancy less than 6 months
18. Concomitant use of strong inhibitors of both cytochrome P450 isoenzyme 3A4 (CYP3A4) and P-glycoprotein (P-gp), i.e., human immunodeficiency virus protease inhibitors and the following azole-antimycotics agents: ketoconazole, itraconazole, voriconazole, or posaconazole, if used systemically
19. Female of childbearing potential who are not surgically sterile, or, if sexually active not willing to use adequate contraceptive measures with a failure rate less than 1% per year (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, male partner sterilization) before entry and throughout the study, as well as pregnant or breast-feeding women
20. Inability to adhere to study procedures
21. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g., employee or student of the investigational site)
22. Previous randomization to this study or participating in a study with an investigational drug or medical device at the time of randomization
23. Antiphospholipid antibody syndrome

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | From randomization to end of recruitment (2 years)
  Recruitment rate of potentially eligible patients from neurology clinics
Refusal rate | From randomization to end of recruitment (2 years)
  Rate of patients who refuse to participate in the clinical trial who otherwise are eligible for the study
Retention rate | From randomization to End of Study (median 2 years)
  Rate of patients who remain in the clinical trial until EOS or qualifying event
Incidence rate of Intracranial hemorrhage | From randomization to End of Study (median 2 years)
  Rate of patients who experience an intracranial hemorrhage during the study

SECONDARY OUTCOMES:
Major hemorrhage | From randomization to End of Study (median 2 years)
  Major hemorrhage as defined by ISTH criteria
Combination of ISTH major hemorrhages & clinically-relevant non-major hemorrhages | From randomization to End of Study (median 2 years)
  Major hemorrhage and clinically relevant non-major as per ISTH criteria
Recurrent ischemic stroke & MRI-detected incident covert brain infarction | From randomization to End of Study (median 2 years)
  Symptomatic investigator reported ischemic stroke and MRI detected covert brain infarct as determined by MRI corelab reading baseline and end of study MRI
Recurrent ischemic stroke | From randomization to End of Study (median 2 years)
  Recurrent ischemic stroke that is restricted to the area of the qualifying stenosis
Composite of stroke, myocardial infarction or vascular death | From randomization to End of Study (median 2 years)
  Composite of stroke, MI or vascular death

CONTACTS AND LOCATIONS:
Overall Officials: Kanjana S. Perera, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (10):
- Canada (10):
  - Alberta Health Services, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Rhema Research Institute, Owen Sound, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perera KS, Sharma MA, Eikelboom JW, Ng KKH, Field TS, Buck BH, Hill MD, Stotts G, Casaubon LK, Mandzia J, Katsanos AH, Yip S, Shoamanesh A, Young GB, Appireddy R, Nayar S, Swartz R, Taylor A, Carrier A, Srivastava A, Deshmukh AS, Zhao R, Hart RG; CATIS-ICAD Investigators. Combination Antithrombotic Therapy for Reduction of Recurrent Ischemic Stroke in Intracranial Atherosclerotic Disease. Stroke. 2025 Feb;56(2):380-389. doi: 10.1161/STROKEAHA.124.047715. Epub 2025 Jan 9. PMID 39781748